CLINICAL TRIAL: NCT01086839
Title: Sino-nasal Inhalation of Sodium Chloride 6,0% in Patients With Cystic Fibrosis and Chronic Rhinosinusitis. A Multicenter, Randomized, Double-blind, Placebo-controlled, Prospective Clinical Trial
Brief Title: Sino-nasal Inhalation of Sodium Chloride 6,0% in Patients With Cystic Fibrosis and Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, PD Dr., University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NaCl 6.0%-nasal-CF
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Cystic Fibrosis; Rhinosinusitis
Keywords: Cystic Fibrosis; chronic rhinosinusitis
MeSH Terms: conditions — Cystic Fibrosis; Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sodium chloride 6% (Experimental): Cross-Over! "experimental" (days 1 - 28), then Wash-Out (28 days),then "placebo comparator" (days 57 - 85).
  Interventions: Drug: sodium chloride 6%
- sodium chloride 0,9% (Placebo Comparator): Cross-Over! "placebo comparator" (days 1 - 28), then Wash-Out (28 days),then "experimental" (days 57 - 85).
  Interventions: Drug: sodium chloride 0,9%

INTERVENTIONS:
Drug: sodium chloride 6% — * one ampoule sodium chloride 6% per day
  * inhalation use
  * for 28 days
  Arms: sodium chloride 6%
Drug: sodium chloride 0,9% — * one ampoule sodium chloride 0,9% per day
  * inhalation use
  * for 28 days
  Arms: sodium chloride 0,9%

SUMMARY:
Rhinosinusitis disorders are almost regularly associated to Cystic Fibrosis (CF). The basic defect in CF is a dysfunction of chloride channels in exocrine glands which equally concerns upper airway mucosa. It leads to retention of secretions and consecutive chronic inflammation with bacterial superinfection.

In CF rhinosinusitis can restrict quality of life, give cause to repeated ear, nose, and throat (ENT) surgery and accelerate disease progression by bacterial acquisition into the airways.

The multicenter, randomized, double-blind, placebo-controlled, prospective clinical trial aims at the evaluation of a sino-nasal inhalation of sodium chloride 6% compared to isotonic saline with respect to ENT-related quality of life which is influenced by mucus retention and the resulting inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of cystic fibrosis based on: 2 positive sweat chloride tests and/or genetic characterization
* Subject is 8 years of age or older
* informed consent of the patient or legal representative
* Women of childbearing potential are only included into the study, if they are using an effective method of birth control during the protocol (failure rate <1% e.g. implants, combined oral contraceptives, injectables, some intrauterine devices, sexual abstinence or vasectomised partner)

Exclusion Criteria:

* Subject has no chronic rhinosinusitis (European Position Paper on Rhinosinusitis and Nasal Polyps (EPOS-criteria)
* Subject has a critical condition defined as: forced expiratory volume at one second < 30% and / or arterial oxygen saturation < 93% without O2-substitution; need of O2-substitution
* Subject had an ENT surgery within 6 months prior to study
* Subject participates in another clinical trial within 30 days prior to study entry

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in the Sino-nasal-outcome test SNOT-20 adapt CF | days 1, 29, 57 and 85

SECONDARY OUTCOMES:
Changes in the nasal lavage fluid and in the serological markers of inflammation | days 1, 29, 57 and 85

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Mainz, M.D., Study Chair — University of Jena
Locations (11):
- Germany (11):
  - Zentrum für Kinder- und Jugendmedizin, Heidelberg, Baden Würtemberg
  - Universitäts-Kinderklinik, Tübingen, Baden-Wurttemberg
  - Medizinische Klinik Innenstadt, München, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Zentrum für Kinder- und Jugendmedizin, Greifswald, Brandenburg
  - J.W. Goethe Universität - Abtl. Pneumologie, Frankfurt am Main, Hesse
  - Klinik für Kinder- und Jugendmedizin, Münster, North Rhine-Westphalia
  - Universitätsklinikum, Leipzig, Saxony
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
  - Mukoviszidosezentrum der Friedrich-Schiller-Universität, Jena, Thuringia
  - CF-Zentrum, Hamburg

REFERENCES:
- [Background] Mainz JG, Koitschev A. Management of chronic rhinosinusitis in CF. J Cyst Fibros. 2009 Jun;8 Suppl 1:S10-4. doi: 10.1016/S1569-1993(09)60005-9. PMID 19460681
- [Background] Mainz JG, Naehrlich L, Schien M, Kading M, Schiller I, Mayr S, Schneider G, Wiedemann B, Wiehlmann L, Cramer N, Pfister W, Kahl BC, Beck JF, Tummler B. Concordant genotype of upper and lower airways P aeruginosa and S aureus isolates in cystic fibrosis. Thorax. 2009 Jun;64(6):535-40. doi: 10.1136/thx.2008.104711. Epub 2009 Mar 11. PMID 19282318
- [Background] Mainz JG, Schien C, Schiller I, Schadlich K, Koitschev A, Koitschev C, Riethmuller J, Graepler-Mainka U, Wiedemann B, Beck JF. Sinonasal inhalation of dornase alfa administered by vibrating aerosol to cystic fibrosis patients: a double-blind placebo-controlled cross-over trial. J Cyst Fibros. 2014 Jul;13(4):461-70. doi: 10.1016/j.jcf.2014.02.005. Epub 2014 Mar 1. PMID 24594542
- [Background] Mainz JG, Schadlich K, Schien C, Michl R, Schelhorn-Neise P, Koitschev A, Koitschev C, Keller PM, Riethmuller J, Wiedemann B, Beck JF. Sinonasal inhalation of tobramycin vibrating aerosol in cystic fibrosis patients with upper airway Pseudomonas aeruginosa colonization: results of a randomized, double-blind, placebo-controlled pilot study. Drug Des Devel Ther. 2014 Feb 10;8:209-17. doi: 10.2147/DDDT.S54064. eCollection 2014. PMID 24596456
- [Derived] Mainz JG, Schumacher U, Schadlich K, Hentschel J, Koitschev C, Koitschev A, Riethmuller J, Prenzel F, Sommerburg O, Wiedemann B, Staab D, Gleiber W, Fischer R, Beck JF, Arnold C; Cooperators. Sino nasal inhalation of isotonic versus hypertonic saline (6.0%) in CF patients with chronic rhinosinusitis - Results of a multicenter, prospective, randomized, double-blind, controlled trial. J Cyst Fibros. 2016 Nov;15(6):e57-e66. doi: 10.1016/j.jcf.2016.05.003. Epub 2016 Jun 5. PMID 27267518